CLINICAL TRIAL: NCT07343791
Title: Efficacy and Safety Study of DC-CIK Cell Therapy Combined With Epaloliposide, Vortexil, and Regorafenib as Third-line Treatment for Advanced Colorectal Cancer.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: JIANG LONGWEI (Other)
Responsible Party: Sponsor-Investigator, JIANG LONGWEI, Associate Researcher, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zlk20251119
Record Dates: First submitted 2025-12-18; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: DC-CIK Treatment; Regorafenib; Colorectal Cancer; Immune Combination Therapy; Iparomlimab and Tuvonralimab Injection
Keywords: DC-CIK treatment; Regorafenib; colorectal cancer; Immune combination therapy; Iparomlimab and Tuvonralimab Injection
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DC-CIK cell immunity combined with Regorafenib,Iparomlimab and Tuvonralimab Injection (Experimental): 1. Epaglitovirizumab: intravenous injection, 5.0 mg/kg, administered on the first day of each 21 day cycle. Continue treatment until disease progression, intolerable toxicity, withdrawal of informed consent, initiation of new anti-tumor therapy, or up to 2 years of use.
  2. Regorafenib: Oral administration, 120mg (3 tablets 40mg), once daily, taken from day 1 to day 21 of a 28 day cycle. Dose adjustment should be made based on patient tolerance, and the minimum dose should not be less than 80mg per day.
  3. DC-CIK cell therapy:
     * Collection and culture: Collect peripheral blood mononuclear cells from patients one day before treatment for in vitro induction and expansion of DC and CIK cells.
     * Return input:
     * DC feedback: 4 times in total. Starting from the 7th day after blood collection, subcutaneous injections were administered in the bilateral inguinal, axillary, and cervical lymph node areas, with a cell count of (1-5) × 10 ^ 7 cells per injection, twice a week.
     * CIK feedback: 3 times i
  Interventions: Combination Product: DC-CIK combined with regorafenib ,Iparomlimab and Tuvonralimab Injection

INTERVENTIONS:
Combination Product: DC-CIK combined with regorafenib ,Iparomlimab and Tuvonralimab Injection — 1. Epaglitovirizumab: intravenous injection, 5.0 mg/kg, administered on the first day of each 21 day cycle. Continue treatment until disease progression, intolerable toxicity, withdrawal of informed consent, initiation of new anti-tumor therapy, or up to 2 years of use.
  2. Regorafenib: Oral administration, 120mg (3 tablets 40mg), once daily, taken from day 1 to day 21 of a 28 day cycle. Dose adjustment should be made based on patient tolerance, and the minimum dose should not be less than 80mg per day.
  3. DC-CIK cell therapy：DC feedback: 4 times in total. Starting from the 7th day after blood collection, subcutaneous injections were administered in the bilateral inguinal, axillary, and cervical lymph node areas, with a cell count of (1-5) × 10 ^ 7 cells per injection, twice a week.
     * CIK feedback: 3 times in total. On the 7th day after blood collection (which may vary by 1-2 days depending on cell growth), intravenous infusion was performed with a cell volu A total of 4 treatment cycles
  Other Names: DC-CIK; regorafenib; Iparomlimab and Tuvonralimab Injection

SUMMARY:
Research background and purpose:

Patients with advanced colorectal cancer face the dilemma of limited treatment options and poor efficacy in the third line treatment stage. Although regorafenib and immune checkpoint inhibitors bring hope to some patients, the efficacy still faces bottlenecks for the vast majority of microsatellite stable patients who are insensitive to immune monotherapy. This study is based on the multi mechanism synergistic theory of "immune activation+vascular inhibition+targeted killing". It innovatively combines autologous DC-CIK cell immunotherapy, domestic PD-1/CTLA-4 bispecific antibody (aparolitovorelli monoclonal antibody), and multi-target tyrosine kinase inhibitor (regorafenib) to evaluate the efficacy and safety of this triple therapy as a third line treatment for advanced colorectal cancer, and explore its immunological mechanism.

Research content and methods:

This study is a single arm, open label clinical trial. Plan to enroll advanced colorectal cancer patients who have previously failed second-line standard treatment. All participants will receive the following combination therapy regimen:

1. Epaglitovirizumab: 5.0 mg/kg, intravenous injection, once every 21 days.
2. Regorafenib: 120mg, once daily, orally, 1-21 days, repeated every 28 days.
3. DC-CIK cell therapy: Collect, culture, and transfuse cells during specific cycles.

The study will strictly follow the protocol for efficacy evaluation (based on RECIST 1.1 standards) and safety monitoring, and a strict quality control and risk management system will be established.

Main evaluation indicators and expected outcomes:

* Primary endpoint: Objective response rate and safety.
* Secondary endpoints: progression free survival, overall survival, duration of remission, and treatment-related immunological responses.
* Expected outcome: This study is expected to provide a promising new comprehensive treatment strategy for chemotherapy resistant advanced colorectal cancer, especially MSS type patients, and break through existing efficacy bottlenecks. The research findings will provide high-level evidence-based medicine for the clinical application of this combined approach and lay the foundation for understanding its synergistic mechanism.

ELIGIBILITY:
Inclusion Criteria:

-1. Sign written informed consent before implementing any experimental procedures; 2. Male or female ≥ 18 years old, ≤ 75 years old; 3. ECOG PS score is 0-1 points; 4. Patients with metastatic colorectal cancer confirmed by histology or cytology; 5. Expected survival time>3 months;

Exclusion Criteria:

-1. It is known that there is active CNS metastasis and/or cancerous meningitis; 2. Chest fluid, ascites, and pericardial effusion that require drainage due to clinical symptoms; 3. Any life-threatening bleeding events that have occurred within the past 3 months, including the need for blood transfusion therapy, surgery or local treatment, and continuous medication therapy; 4. Uncontrollable hypertension, with systolic blood pressure>150mmHg or diastolic blood pressure>90 mmHg after optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy; 5. Human immunodeficiency virus (HIV) infected individuals (HIV 1/2 antibody positive), known syphilis infected individuals;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS)- Evaluate the effectiveness of DC-CIK cell therapy combined with aparolitovorelizumab and regorafenib regimen as a third line therapy in patients with advanced colorectal cancer. | From enrollment to the end of treatment (2 years)
  The efficacy effectiveness are evaluated by progression free survival (PFS)
objective clinical response using RESIST(version 1.1) | From enrollment to the end of treatment (2 years)
  Evaluate the effectiveness of DC-CIK cell therapy combined with aparolitovorelizumab and regorafenib regimen as a third line therapy in patients with advanced colorectal cancer.

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of the combination therapy. | From enrollment to the end of the study (2 years)
  Safety and tolerability were evaluated using Common Terminology Criteria for Adverse Events (CTCAE 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zengjie, Study Chair — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No